CLINICAL TRIAL: NCT02158728
Title: Supraventricular Tachycardia Collection Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: SVT Collect Study
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Supraventricular Arrhythmias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD indicated subjects: Subjects indicated for implantable cardioverter defibrillator (ICD)/ cardiac resynchronization therapy defibrillator (CRT-D) implant, ICD/CRT-D change-out, or indicated for an ICD/CRT-D and undergoing ablation or electrophysiology (EP) study (including Non-Invasive ElectroPhysiology Study [NIPS]).
  Enrolled subjects are prepared for the indicated procedure as per investigational center's standard practice. The investigator will determine the best methodology for inducing or simulating SVT within the indicated procedure. Data is recorded by a data acquisition recording system. Recording should begin just before the indicated procedure and continue until completion of the procedure.The recorded data are collected.

SUMMARY:
To collect supraventricular tachycardia (SVT) data for developing and testing sensing and detection algorithms for a subcutaneous implantable cardioverter defibrillator (ICD).

DETAILED DESCRIPTION:
The purpose of the SVT Collect study is to collect supraventricular tachycardia episode data for developing and testing new sensing and detection algorithms for a future subcutaneous ICD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or above, or of legal age to give consent specific to the national law of the countries in which the trial is being conducted
* Subjects indicated for implantable cardioverter defibrillator (ICD)/cardiac resynchronization therapy defibrillator (CRT-D) implant or ICD/CRT-D change-out, OR subjects indicated for an ICD/CRT-D that are undergoing ablation or electrophysiology (EP) study (including Non-invasive EP Study [NIPS])
* Subjects are willing to provide Informed Consent

Exclusion Criteria:

* Subjects who are ventricular pacing dependent
* Subjects with a preexisting dual/triple chamber pacemaker or ICD who have a history of atrioventricular (AV) block with atrial pacing < 120 beats per minute (BPM) while awake.
* Subjects who are unable to tolerate elevated ventricular rates (≥170BPM)
* Any condition which precludes the subject's ability to comply with the study requirements
* Enrollment in a concurrent study (without prior study management approval) that may confound the results of this study
* Subjects who are legally incompetent
* Subjects meet exclusion criteria required by local laws and regulations (e.g. age, breast feeding, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Implantable cardioverter defibrillator (ICD) indicated
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ICD Indicated Subjects: Subjects indicated for ICD/CRT-D implant, ICD/CRT-D change-out, or indicated for an ICD/CRT-D and undergoing ablation or electrophysiology (EP) study (including Non-invasive EP study [NIPS])
  ICD: implantable cardioverter defibrillator CRT-D: cardiac resynchronization therapy defibrillator
Period: Overall Study
Arm/Group | ICD Indicated Subjects
Started | 80
Completed | 53
Not Completed | 27
Not completed — no procedure according to CIP done | 3
Not completed — no qualified dataset | 24

BASELINE CHARACTERISTICS:
Population: ICD-indicated subjects undergoing standard ICD/CRT-D implant, ICD/CRT-D change-out, ablation, electrophysiology (EP) study or Non Invasive Programmed Stimulation (NIPS), and who provided a dataset which qualified for developing and testing the sensing and detection algorithms of the new ICD, are included in the analyses.
Groups:
- ICD Indicated Subjects: Subjects indicated for implantable cardioverter defibrillator (ICD)/cardiac resynchronization therapy defibrillator (CRT-D) implant, ICD/CRT-D change-out, or indicated for an ICD/CRT-D and undergoing ablation or electrophysiology (EP) study (including Non-Invasive ElectroPhysiology Study [NIPS]).
Arm/Group | ICD Indicated Subjects
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 37
Region of Enrollment [Number; unit: participants]
  Hungary | 6
  Taiwan | 21
  Hong Kong | 11
  Slovakia | 13
  China | 2
Indication for implantable cardioverter defibrillator (ICD) [Number; unit: participants] | 47
Indication for cardiac resynchronization therapy defibrillator (CRT-D) [Number; unit: participants] | 6
Hypertension [Number; unit: participants] | 25
Congestive Heart Failure [Number; unit: participants] | 31
Coronary Artery Disease [Number; unit: participants] | 24
Previous myocardial infarction [Number; unit: participants] | 17
Sinus atrioventricular (AV) junctional arrhythmias and blocks [Number; unit: participants] | 23
Sinus arrhythmias [Number; unit: participants] | 13
Atrial arrhythmias [Number; unit: participants] | 15
Ventricular arrhythmias [Number; unit: participants] | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Electrocardiograms (ECGs) Collected
Description: Collected were the number of ECGs received from the enrolled subjects, the number of ECGs with SVT (supraventricular tachycardia) episodes, and the number of ECGs with SVT episodes qualified for algorithm development and validation of the potential new ICD. The ECG data were collected continuously during the indicated procedure (ICD/CRT-D implant, ICD/CRT-D change-out, electrophysiology (EP) study (including non invasive EP study)
Time Frame: After recorded ECGs had been received, which were collected until the end of the indicated procedure
Population: Total number of ECGs received from the 80 enrolled subjects.
Measure: Number; unit: ECG
Groups:
- ICD Indicated Subjects: From the initially 80 enrolled subjects indicated for ICD/CRT-D implant, ICD/CRT-D change-out, or indicated for an ICD/CRT-D and undergoing ablation or EP study (including Non-invasive EP Study [NIPS]), 53 subjects provided SVT episode data which qualified for developing and testing new sensing and detection algorithms for a new MedtronicICD. SVT episodes with a ventricular response rate of ≥170 BPM are required in the development of the algorithms.
Arm/Group | ICD Indicated Subjects
Number analyzed (Participants) | 80
ECG
  Number of ECGs received | 77
  Number of ECGs with SVT episodes | 67
  Number of ECGs with qualified SVT episodes | 53

ADVERSE EVENTS:
Time Frame: From the first enrolled patient until the last exited patient. Which is from June 11, 2014 up to October 27, 2015
Groups:
- ICD Indicated Subjects: Only ICD-indicated subjects undergoing standard ICD/CRT-D implant, ICD/CRT-D change-out, ablation, electrophysiology (EP) study or Non Invasive Programmed Stimulation (NIPS), and who provided a dataset which qualified for developing and testing the sensing and detection algorithms of the new ICD, are included in the analyses.
Arm/Group | ICD Indicated Subjects
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No